CLINICAL TRIAL: NCT07288372
Title: An Exploratory Investigation Into the Mechanism of Glycemic Homeostasis Regulation Under the Synergistic Conditions of Continuous Glucose Monitoring (CGM) and Oral Glucose Tolerance Test (OGTT)
Brief Title: The CGM-OGTT Glycemic Homeostasis Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Principal Investigator, Professor, Chief Physician, Head of Department, Shanghai 6th People's Hospital
Other Study IDs: 20251120
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Glucose Metabolism Disorders
Keywords: Continuous Glucose Monitoring; CGM; Oral Glucose Tolerance Test; OGTT; Mixed-Meal Tolerance Test; Glycemic Variability; Incretins; Home-Based Testing; GLP-1; GIP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Glucose Tolerance (NGT): Participants with normal glucose tolerance as defined by a 2-hour plasma glucose value < 7.8 mmol/L during the oral glucose tolerance test (OGTT).
- Pre-diabetes (Pre-DM): Participants with pre-diabetes (intermediate hyperglycemia) as defined by a 2-hour plasma glucose value between 7.8 mmol/L and 11.0 mmol/L during the OGTT.
- Newly Diagnosed Type 2 Diabetes (T2DM): Participants with newly diagnosed type 2 diabetes as defined by a 2-hour plasma glucose value ≥ 11.1 mmol/L during the OGTT.

SUMMARY:
This is a prospective, exploratory, observational study aimed at investigating the mechanisms of glycemic homeostasis by comparing continuous glucose monitoring (CGM) data with results from the oral glucose tolerance test (OGTT).

The study plans to enroll approximately 225 participants aged 18-70 years who are at risk for or suspected of having glucose metabolism disorders, but without a prior diagnosis of diabetes. Participants will be equipped with a blinded CGM device for 10-14 days. During this period, they will perform two standardized mixed-meal tolerance tests (MMTT) at home. Subsequently, they will undergo a standard 75g OGTT at the hospital, where blood samples will be collected at multiple time points to measure glucose, insulin, C-peptide, and gastrointestinal hormones (GLP-1, GIP).

Based on the 2-hour blood glucose value from the OGTT, participants will be naturally categorized into three groups for comparative analysis: Normal Glucose Tolerance (NGT), Pre-diabetes (Pre-DM), and Newly Diagnosed Type 2 Diabetes (T2DM).

The primary objective is to establish a quantitative relationship between CGM-derived parameters (e.g., glycemic variability, time-in-range) after the MMTT and the OGTT diagnostic results. Secondary objectives include assessing the feasibility and correlation between home-based MMTT and standard OGTT, exploring the impact of gastrointestinal hormone responses on daily glucose fluctuations, and investigating the association between postprandial glucose dynamics and vascular reactivity (e.g., postprandial hypotension).

DETAILED DESCRIPTION:
Background and Rationale:

The oral glucose tolerance test (OGTT) is the gold standard for diagnosing diabetes but has limitations, including its inability to reflect daily glycemic variability and the discomfort caused by a high glucose load, which may not represent physiological conditions. Continuous glucose monitoring (CGM) captures comprehensive glycemic fluctuations in free-living settings. The mixed-meal tolerance test (MMTT), containing macronutrients like fat and protein, better simulates a physiological meal and may be better tolerated. However, the quantitative relationship between CGM-derived parameters from home-based MMTTs and the diagnostic outcomes of the standard OGTT remains unclear. Furthermore, the role of gastrointestinal hormone responses (e.g., GLP-1, GIP) during an OGTT in modulating subsequent daily glycemic homeostasis is an area of exploratory interest. This study aims to bridge these gaps by synergistically utilizing CGM, MMTT, and OGTT to investigate the mechanisms of glycemic regulation.

Study Design and Methodology:

This is a single-center, prospective, exploratory, observational study. Participants will wear a blinded CGM sensor for 10-14 days to prevent behavioral bias. The study comprises three sequential phases:

At-home MMTT Phase (Day 2 and another day prior to hospital visit): Participants will perform two standardized MMTTs (a standard formula and a high-protein formula) at home after an overnight fast. Adherence and any adverse events will be monitored remotely via a dedicated mini-program and daily communication.

In-hospital OGTT and Biomarker Assessment Phase (Day 10-14): Participants will undergo a standard 75g OGTT at the clinic. Venous blood samples will be collected at fasting, 30, 60, 120, and 180 minutes for measuring glucose, insulin, C-peptide, GLP-1, GIP, and blood pressure/heart rate.

Group Allocation:

This is an observational study with no interventional allocation. After completion, participants will be categorized into three groups based solely on their 2-hour plasma glucose (2hPG) value from the OGTT, following WHO criteria: Normal Glucose Tolerance (NGT, 2hPG <7.8 mmol/L), Pre-diabetes (Pre-DM, 7.8 ≤ 2hPG <11.1 mmol/L), and Type 2 Diabetes (T2DM, 2hPG ≥11.1 mmol/L). Comparative analyses will be conducted across these naturally formed groups.

Statistical Considerations:

The sample size of 225 was calculated using G*Power for an ANOVA model (effect size f=0.25, α=0.05, power=0.80), accounting for a 20% dropout rate. The primary analysis will use the Full Analysis Set (FAS). Statistical methods will include Spearman correlation to assess the relationship between MMTT-induced CGM parameters and OGTT glucose values, Analysis of Covariance (ANCOVA) to compare CGM metrics across the three glycemic groups (adjusting for covariates like age and BMI), and Receiver Operating Characteristic (ROC) curve analysis to evaluate the predictive power of CGM parameters for OGTT-based diagnosis.

Scientific Value:

This study is designed as a mechanism-exploratory investigation. It seeks to validate a novel, patient-centric approach (home-based MMTT with CGM) against the diagnostic gold standard (OGTT) and to provide deeper insights into the integrated physiology of glycemic homeostasis, including the role of incretin hormones and its potential link to vascular responses like postprandial hypotension.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet ALL of the following criteria:

* Is aged between 18 and 70 years, inclusive.
* And meets at least ONE of the following conditions:

  * Presents with diabetes-related clinical symptoms or signs (e.g., unexplained ·polydipsia, polyphagia, polyuria, weight loss) and has been advised by a ·clinician to undergo an OGTT for diagnostic clarification.
  * Has indicators of abnormal glucose metabolism:Impaired Fasting Glucose (IFG): Fasting venous plasma glucose ≥ 6.1 mmol/L and < 7.0 mmol/L.and/or Glycated hemoglobin (HbA1c) in the pre-diabetes range of 5.7% to 6.4%.
  * Has at least one of the following diabetes risk factors:Body Mass Index (BMI) ≥ 24 kg/m²；Has a first-degree relative (parent, sibling, or child) with a history of diabetes；Has a history of hypertension (or undergoing antihypertensive treatment) or dyslipidemia.

Exclusion Criteria:

* An individual who meets ANY of the following criteria will be excluded from participation in this study:
* Previously diagnosed with diabetes.
* Use of medications that significantly affect glucose metabolism or gastrointestinal hormones (e.g., GLP-1 receptor agonists, DPP-4 inhibitors, glucocorticoids) within a specified washout period prior to enrollment.
* History of gastrointestinal surgery (e.g., gastrectomy) or chronic pancreatic disease.
* Presence of severe hepatic or renal impairment (e.g., ALT > 3 times the upper limit of normal, or eGFR < 45 mL/min/1.73m²).
* Pregnant or lactating women, or women planning to become pregnant during the study period.
* Known allergy to soy (as the standardized meal may contain soy-based components).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This monocentric, prospective, observational study will enroll 225 adult participants (aged 18-70 years) who are at high risk for diabetes or present with abnormal glucose metabolism, but have not been previously diagnosed with diabetes.
  Participants must meet specific eligibility criteria, including having diabetes-related symptoms, impaired fasting glucose, elevated HbA1c in the pre-diabetes range, or established risk factors (e.g., obesity, family history of diabetes, hypertension, or dyslipidemia).
  Key Exclusion Criteria include a prior diagnosis of diabetes, use of medications affecting glucose metabolism, significant organ dysfunction, or pregnancy.
  Upon enrollment, all participants will undergo a standardized 75g Oral Glucose Tolerance Test (OGTT). Based on the OGTT results, they will be retrospectively categorized into three natural groups for comparative analysis: Normal Glucose Tolerance (NGT), Pre-Diabetes (Pre-DM), and Newly Diagnosed Type 2 Diabetes (T2DM).
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between MMTT-induced glucose AUC and OGTT plasma glucose values | MMTT: 0-3 hours post-meal (for AUC calculation). OGTT: 0, 30, 60, 120, and 180 minutes (for plasma glucose values).
  To establish a quantitative relationship by assessing the correlation between the area under the curve (AUC) of postprandial glucose derived from Continuous Glucose Monitoring (CGM) after a standardized Mixed-Meal Tolerance Test (MMTT) and the plasma glucose values at all standard time points during the Oral Glucose Tolerance Test (OGTT).

SECONDARY OUTCOMES:
Glycemic Variability (GV) | Entire CGM monitoring period (10-14 days)
  Coefficient of variation (CV) of glucose levels, calculated from Continuous Glucose Monitoring (CGM) data.
Dietary Macronutrient Intake Composition | From enrollment until the completion of the in-clinic OGTT (approximately 10-14 days).
  The daily intake proportion of macronutrients (carbohydrates, protein, and fat), expressed as a percentage of total caloric intake, assessed via a dietary logging application.
Caloric Intake per Meal | From enrollment until the completion of the in-clinic OGTT (approximately 10-14 days).
  The average energy intake (in kilocalories) per meal, estimated using a dietary logging application.
Mean Amplitude of Glycemic Excursions (MAGE) | Entire CGM monitoring period (10-14 days)
  Mean Amplitude of Glycemic Excursions, calculated from CGM data to quantify major glucose swings.
Complexity of Glucose Time Series | Entire CGM monitoring period (10-14 days)
  Complexity of glucose time series (e.g., using multiscale entropy or similar indices) derived from CGM data.
Glucose AUC after MMTT | 0-3 hours after each MMTT
  Area under the curve of glucose levels after each Mixed-Meal Tolerance Test (MMTT), measured by CGM.
Glucose Levels During OGTT | OGTT: 0, 30, 60, 120, 180 minutes
  Plasma levels of glucose at OGTT time points
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline (OGTT 0-minute sample)
  Insulin resistance index calculated from fasting glucose and fasting insulin levels.
Incidence of Postprandial Hypotension during OGTT | OGTT: 0, 30, 60, 120, 180 minutes
  Occurrence of postprandial hypotension, defined as a maximum decrease in systolic blood pressure ≥ 20 mmHg from baseline after the OGTT.
Maximum reduction in systolic blood pressure (SBP) during OGTT | OGTT: 0, 30, 60, 120, 180 minutes
  The maximum decrease (Δ) in systolic blood pressure from the baseline (pre-glucose ingestion) value at any standard time point during the Oral Glucose Tolerance Test.
Completion Rate of Home-based MMTT | Through study completion (up to 14 days)
  Proportion of participants who successfully complete both home-based MMTTs.
Adverse Events during OGTT /MMTT | During the OGTT/MMTT procedure (approximately 3 hours)
  Incidence of adverse events (e.g., nausea, vomiting, bloating) occurring during the OGTT/MMTT procedure.
GLP-1 serum concentration during OGTT | OGTT: 0, 30, 60, 120, and 180 minutes
  Serum concentration of Glucagon-like peptide-1 (GLP-1) at each standard time point in response to the Oral Glucose Tolerance Test (OGTT).
GIP serum concentration during OGTT | OGTT: 0, 30, 60, 120, and 180 minutes
  Serum concentration of Glucose-dependent insulinotropic polypeptide (GIP) at each standard time point in response to the Oral Glucose Tolerance Test (OGTT).
Insulin serum concentration during OGTT | OGTT: 0, 30, 60, 120, 180 minutes
  Plasma insulin concentration at each time point of the Oral Glucose Tolerance Test (OGTT).
C-peptide serum concentration during OGTT | OGTT: 0, 30, 60, 120, 180 minutes
  Plasma C-peptide concentration at each time point of the Oral Glucose Tolerance Test (OGTT).
Total GLP-1 AUC during OGTT | OGTT: 0, 30, 60, 120, and 180 minutes
  Total area under the curve (AUC) for the Glucagon-like peptide-1 (GLP-1) serum concentration profile in response to the Oral Glucose Tolerance Test (OGTT).
Total GIP AUC during OGTT | OGTT: 0, 30, 60, 120, and 180 minutes
  Total area under the curve (AUC) for the Glucose-dependent insulinotropic polypeptide (GIP) serum concentration profile in response to the Oral Glucose Tolerance Test (OGTT).
Association between Incretin Secretion and Glycemic Complexity | During the in-clinic OGTT （0 to 180 minutes）
  An exploratory analysis using multiple linear regression to assess the influence of GLP-1 AUC and GIP AUC (during OGTT) on the complexity of the glycemic time series (e.g., CGI) during the OGTT period, adjusting for covariates such as age, sex, and BMI.
Time to Peak Glucose after Each Meal | Throughout the CGM monitoring period (10-14 days), following each main meal.
  The time (in minutes) from the start of a meal to the maximum postprandial glucose concentration, as determined by CGM data. The average for breakfast, lunch, and dinner will be calculated.
Maximum reduction in diastolic blood pressure (DBP) during OGTT | OGTT: 0, 30, 60, 120, and 180 minutes
  The maximum decrease (Δ) in diastolic blood pressure from the baseline (pre-glucose ingestion) value at any standard time point during the Oral Glucose Tolerance Test.
Glycated hemoglobin (HbA1c) level | OGTT day (single time point, e.g., at the fasting blood draw)
  The concentration of glycated hemoglobin (HbA1c) in venous blood samples collected on the day of the Oral Glucose Tolerance Test (OGTT). HbA1c reflects the average blood glucose level over the preceding 2 to 3 months
Glycated albumin (GA) level | OGTT day (single time point, e.g., at the fasting blood draw)
  The concentration of glycated albumin (GA) in venous blood samples collected on the day of the Oral Glucose Tolerance Test (OGTT). GA reflects the average blood glucose level over the preceding 2 to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Study Chair — Shanghai Sixth People's Hospital, Shanghai, Shanghai 200233

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study are highly sensitive, containing detailed glycemic profiles, hormone levels, and personal health information. To protect participant confidentiality and privacy as strictly stipulated in the informed consent form and approved by the ethics committee, the IPD will not be made publicly available. The data will be de-identified and stored securely for analysis by the principal investigative team only. In the future, requests for access to anonymized data may be considered on a case-by-case basis for legitimate scientific collaboration, subject to a formal data sharing agreement and approval from the institutional ethics committee.